CLINICAL TRIAL: NCT05917782
Title: A Randomized, Open-Label, Parallel-Designed, Phase I Clinical Study to Evaluate the Pharmacokinetics Similarity of Single-Dose CBP-201 Injection With Different Dosage Forms and Strengths in Healthy Adult Chinese Subjects
Brief Title: A Study to Evaluate the Pharmacokinetics Similarity of CBP-201 in Healthy Adult Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Connect Biopharm LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CBP-201-CN004
Record Dates: First submitted 2023-06-04; First posted 2023-06-26 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Healthy Adult Subjects
MeSH Terms: interventions — Drug Evaluation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test drug (T1): CBP-201 injection (pre-filled syringe, 150 mg/1 mL) (Experimental): Strength: pre-filled syringe, 150 mg/1 mL
  Interventions: Biological: Test drug (T1): CBP-201 injection (pre-filled syringe, 150 mg/1 mL)
- Test drug (T2): CBP-201 injection (pre-filled syringe, 300 mg/2 mL) (Experimental): Strength: pre-filled syringe, 300 mg/2 mL
  Interventions: Biological: Test drug (T2): CBP-201 injection (pre-filled syringe, 300 mg/2 mL)
- Reference drug (R): CBP-201 injection (vial, 150 mg/1 mL) (Active Comparator): Strength: vial, 150 mg/1 mL
  Interventions: Biological: Reference drug (R): CBP-201 injection (vial, 150 mg/1 mL)

INTERVENTIONS:
Biological: Test drug (T1): CBP-201 injection (pre-filled syringe, 150 mg/1 mL) — subcutaneous injection of 2 doses on Day 1
  Arms: Test drug (T1): CBP-201 injection (pre-filled syringe, 150 mg/1 mL)
Biological: Test drug (T2): CBP-201 injection (pre-filled syringe, 300 mg/2 mL) — subcutaneous injection of 1 dose on Day 1
  Arms: Test drug (T2): CBP-201 injection (pre-filled syringe, 300 mg/2 mL)
Biological: Reference drug (R): CBP-201 injection (vial, 150 mg/1 mL) — subcutaneous injection of 2 doses on Day 1
  Arms: Reference drug (R): CBP-201 injection (vial, 150 mg/1 mL)

SUMMARY:
This is a single-center, randomized, open-label, single-dose, parallel-designed PK similarity study.

DETAILED DESCRIPTION:
A total of 324 healthy subjects are planned to be enrolled and randomized into 3 groups at a ratio of 1:1:1, with 108 subjects in each group. They will receive 2 doses of the test drug T1 (CBP-201 injection (pre-filled syringe, 150 mg/1 mL)), 1 dose of the test drug T2 (CBP-201 injection (pre-filled syringe, 300 mg/2 mL)), and 2 doses of the reference drug R (CBP-201 injection (vial, 150 mg/1 mL)), respectively.

The study consists of a screening period (Day-28 to Day-2), a baseline period (Day-1), an administration and observation period (Day1 to Day6), and a follow-up period (Day7 to Day57).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are to read, understand, and sign the ICF.
2. Healthy adult male or female subjects aged 18-45 years (inclusive) at screening, with each sex accounting for at least one-third of the overall sample size.
3. Body mass index (BMI) is between 19 and 28 kg/m2 (inclusive). Male subjects weigh ≥ 50 kg, and female subjects weigh ≥ 45 kg.
4. Subjects with partners must agree to take medically accepted effective contraceptive measures (including physical contraception, surgery, abstinence, etc) from signing of the ICF until 90 days after administration.
5. The results of vital sign assessment, physical examination, clinical laboratory tests (hematology, urinalysis, biochemistry, coagulation) and 12-lead ECG at screening or baseline are normal or abnormal but not clinically significant.
6. Subjects who are able to communicate well with the clinical staff and complete the study according to the protocol.

Exclusion Criteria:

1. Subjects who have diseases or conditions with abnormal clinical manifestations, including but not limited to renal, cardiac, hematological, bronchial, pulmonary, vascular, gastrointestinal, allergic, neurological, endocrine and metabolic diseases (diabetes mellitus, thyroid disorder, and adrenal disorder), skeletal disease and immunodeficiency, cancer, and hepatitis, or cirrhosis.
2. Subjects with allergic diseases (such as allergic rhinitis, allergic asthma) at screening, a history of systemic anaphylaxis, or who may be allergic to any component of the test drugs or similar drugs as determined by the investigator.
3. Subjects who have donated blood or have had substantial loss of blood (> 400 mL) within 3 months before administration.
4. Subjects who have been vaccinated with live (attenuated) vaccines within 3 months before administration.
5. Subjects who have participated in clinical studies of other drugs within 3 months before administration.
6. Subjects who have taken any prescription drugs, over-the-counter drugs, vitamin products, Chinese patent medicines, and Chinese herbal medicines within 1 month before administration.
7. Subjects who have been diagnosed with clinically significant diseases or have undergone major surgical procedures within 1 month before administration, or who are scheduled to undergo major surgery during the study.
8. Female subjects who test positive for pregnancy at screening or baseline or who are lactating.
9. Subjects who smoke more than 5 cigarettes or equivalent per day within 3 months before administration.
10. Subjects who have a history of drug abuse within the last 5 years, who have used narcotics within 3 months before administration, or who test positive in urine drug screening at the screening/baseline visit.
11. Subjects who have a history of regular alcohol consumption, which is defined as consumption of more than 7 units of alcohol per week for females or more than 14 units of alcohol per week for males (1 unit of alcohol equals 360 mL of beer, 45 mL of 40% liquor, or 150 mL of wine) within 3 months before administration, who take any alcohol-containing product within 48 h before administration, or who test positive in blood alcohol tests at the screening/ baseline visit.
12. Subjects with known symptoms of dermatitis or skin abnormalities at and around the site of administration.
13. Subjects who test positive for treponema pallidum antibody (TP-Ab), hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb) or hepatitis C virus antibody (HCV-Ab), and human immunodeficiency virus antibody (HIV-Ab).
14. Patients with active tuberculosis, latent tuberculosis, or nontuberculous mycobacterial infection at screening;

    Notes:
    * Unless treatment records clearly documented by a specialist demonstrate that the patients have been adequately treated and may begin treatment with biological product (based on the medical judgment by the investigator and/or infectious disease specialist);
    * If needed, T-spot tests may be used to assist diagnosis of suspected tuberculosis.
15. Subjects with white blood cell count and neutrophil count below the lower limit of normal.
16. Female subjects with hemoglobin values less than 110 g/L or male subjects less than 120 g/L.
17. Subjects who cannot tolerate venous blood sampling, or who have a history of acupuncture syncope or hemophobia.
18. Subjects who still need or plan to engage in strenuous physical activity or exercise during the study.
19. Any other conditions that the investigator determines may affect the subject's provision of informed consent or compliance with the study protocol, or that the investigator deems unsuitable for participation in this study, or the subjects' participation in the study may affect the study results or their own safety.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 324 (Actual)
Dates: Start 2023-07-18 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2023-10-06 (Actual)

PRIMARY OUTCOMES:
Cmax: Maximum concentration | Pre-dose and 6hour, 24hour, 48hour, 72hour, 96hour, 120hour, Day8, Day10, Day11, Day12, Day15, Day18, Day22, Day29, Day36, Day43, Day57 post-dose
  Pharmacokinetics similarity evaluation for test drug T1, test drug T2 and reference drug R
AUC0-t: Area under the plasma concentration-time curve from the start of administration to the last measurable concentration time point T | Pre-dose and 6hour, 24hour, 48hour, 72hour, 96hour, 120hour, Day8, Day10, Day11, Day12, Day15, Day18, Day22, Day29, Day36, Day43, Day57 post-dose
  Pharmacokinetics similarity evaluation for test drug T1, test drug T2 and reference drug R
AUC0-inf: Area under the plasma concentration-time curve from the start of administration to infinity | Pre-dose and 6hour, 24hour, 48hour, 72hour, 96hour, 120hour, Day8, Day10, Day11, Day12, Day15, Day18, Day22, Day29, Day36, Day43, Day57 post-dose
  Pharmacokinetics similarity evaluation for test drug T1, test drug T2 and reference drug R

SECONDARY OUTCOMES:
Maximum concentration (Cmax) | Pre-dose and 6hour, 24hour, 48hour, 72hour, 96hour, 120hour, Day8, Day10, Day11, Day12, Day15, Day18, Day22, Day29, Day36, Day43, Day57 post-dose
  Calculated by non-compartmental analysis (NCA) using WinNonLin V8.3.1 (or higher version)
Area under the plasma concentration-time curve from the start of administration to the last measurable concentration time point T (AUC0-t) | Pre-dose and 6hour, 24hour, 48hour, 72hour, 96hour, 120hour, Day8, Day10, Day11, Day12, Day15, Day18, Day22, Day29, Day36, Day43, Day57 post-dose
  Calculated by non-compartmental analysis (NCA) using WinNonLin V8.3.1 (or higher version)
Area under the plasma concentration-time curve from the start of administration to infinity (AUC0-inf) | Pre-dose and 6hour, 24hour, 48hour, 72hour, 96hour, 120hour, Day8, Day10, Day11, Day12, Day15, Day18, Day22, Day29, Day36, Day43, Day57 post-dose
  Calculated by non-compartmental analysis (NCA) using WinNonLin V8.3.1 (or higher version)
Time to peak (Tmax) | Pre-dose and 6hour, 24hour, 48hour, 72hour, 96hour, 120hour, Day8, Day10, Day11, Day12, Day15, Day18, Day22, Day29, Day36, Day43, Day57 post-dose
  Calculated by non-compartmental analysis (NCA) using WinNonLin V8.3.1 (or higher version)
Elimination half-life (t1/2) | Pre-dose and 6hour, 24hour, 48hour, 72hour, 96hour, 120hour, Day8, Day10, Day11, Day12, Day15, Day18, Day22, Day29, Day36, Day43, Day57 post-dose
  Calculated by non-compartmental analysis (NCA) using WinNonLin V8.3.1 (or higher version)
Apparent clearance (CL/F) | Pre-dose and 6hour, 24hour, 48hour, 72hour, 96hour, 120hour, Day8, Day10, Day11, Day12, Day15, Day18, Day22, Day29, Day36, Day43, Day57 post-dose
  Calculated by non-compartmental analysis (NCA) using WinNonLin V8.3.1 (or higher version)
Apparent volume of distribution (Vz/F) | Pre-dose and 6hour, 24hour, 48hour, 72hour, 96hour, 120hour, Day8, Day10, Day11, Day12, Day15, Day18, Day22, Day29, Day36, Day43, Day57 post-dose
  Calculated by non-compartmental analysis (NCA) using WinNonLin V8.3.1 (or higher version)
Terminal elimination phase rate constant (λz) | Pre-dose and 6hour, 24hour, 48hour, 72hour, 96hour, 120hour, Day8, Day10, Day11, Day12, Day15, Day18, Day22, Day29, Day36, Day43, Day57 post-dose
  Calculated by non-compartmental analysis (NCA) using WinNonLin V8.3.1 (or higher version)
Adverse events (AEs) | Up to 57 days post dosing
  All adverse events will be coded using Medical Dictionary for Regulatory Activities (MedDRA) (the latest version).
Injection site reactions | Day1, Day2, Day3, Day4, Day6, Day8, Day15, Day22, Day29, Day57
  The injection site will be examined and the results will be judged by the investigator.
Blood Pressure (systolic and diastolic blood pressures) | pre-dose, Day1, Day2, Day3, Day4, Day6, Day8, Day10, Day11, Day12, Day15, Day18, Day22, Day29, Day36, Day43, Day57
  The results as well as their changes from baseline will be statistically summarized by dose group and visit.
Pulse | pre-dose, Day1, Day2, Day3, Day4, Day6, Day8, Day10, Day11, Day12, Day15, Day18, Day22, Day29, Day36, Day43, Day57
  The results as well as their changes from baseline will be statistically summarized by dose group and visit.
Body Temperature (ear temperature) | pre-dose, Day1, Day2, Day3, Day4, Day6, Day8, Day10, Day11, Day12, Day15, Day18, Day22, Day29, Day36, Day43, Day57
  The results as well as their changes from baseline will be statistically summarized by dose group and visit.
Respiratory Rate | pre-dose, Day1, Day2, Day3, Day4, Day6, Day8, Day10, Day11, Day12, Day15, Day18, Day22, Day29, Day36, Day43, Day57
  The results as well as their changes from baseline will be statistically summarized by dose group and visit.
Physical examination | pre-dose, Day6, Day15, Day29, Day57
  Physical examination items include: skin (including observation of the planned injection site (abdomen) and surrounding skin during the screening period and at baseline), lymph nodes, head, eyes, neck, chest, abdomen, spine/extremities, and nervous system. The results of physical examination will be evaluated by investigator's observation.
12-lead electrocardiogram (ECG) | pre-dose, Day1, Day2, Day4, Day6, Day10, Day15, Day22, Day29, Day36, Day43, Day57
  ECG variables include ventricular heart rate, PR interval, QRS interval, QT interval, and QTcF interval.
Clinical laboratory test: Hematology - Hemoglobin (Hgb) | pre-dose, Day6, Day15, Day29, Day43, Day57
  The results of clinical laboratory tests, as well as their changes from baseline will be statistically summarized by dose group and visit.
Clinical laboratory test: Hematology - Hematocrit (Hct) | pre-dose, Day6, Day15, Day29, Day43, Day57
  The results of clinical laboratory tests, as well as their changes from baseline will be statistically summarized by dose group and visit.
Clinical laboratory test: Hematology - red blood cell count (RBC) | pre-dose, Day6, Day15, Day29, Day43, Day57
  The results of clinical laboratory tests, as well as their changes from baseline will be statistically summarized by dose group and visit.
Clinical laboratory test: Hematology - platelet count | pre-dose, Day6, Day15, Day29, Day43, Day57
  The results of clinical laboratory tests, as well as their changes from baseline will be statistically summarized by dose group and visit.
Clinical laboratory test: Hematology - white blood cell count (WBC) | pre-dose, Day6, Day15, Day29, Day43, Day57
  The results of clinical laboratory tests, as well as their changes from baseline will be statistically summarized by dose group and visit.
Clinical laboratory test: Hematology - lymphocyte count | pre-dose, Day6, Day15, Day29, Day43, Day57
  The results of clinical laboratory tests, as well as their changes from baseline will be statistically summarized by dose group and visit.
Clinical laboratory test: Hematology - lymphocyte percentage | pre-dose, Day6, Day15, Day29, Day43, Day57
  The results of clinical laboratory tests, as well as their changes from baseline will be statistically summarized by dose group and visit.
Clinical laboratory test: Hematology - neutrophil count | pre-dose, Day6, Day15, Day29, Day43, Day57
  The results of clinical laboratory tests, as well as their changes from baseline will be statistically summarized by dose group and visit.
Clinical laboratory test: Hematology - neutrophil percentage | pre-dose, Day6, Day15, Day29, Day43, Day57
  The results of clinical laboratory tests, as well as their changes from baseline will be statistically summarized by dose group and visit.
Clinical laboratory test: Hematology - monocyte count | pre-dose, Day6, Day15, Day29, Day43, Day57
  The results of clinical laboratory tests, as well as their changes from baseline will be statistically summarized by dose group and visit.
Clinical laboratory test: Hematology - monocyte percentage | pre-dose, Day6, Day15, Day29, Day43, Day57
  The results of clinical laboratory tests, as well as their changes from baseline will be statistically summarized by dose group and visit.
Clinical laboratory test: Hematology - eosinophil count | pre-dose, Day6, Day15, Day29, Day43, Day57
  The results of clinical laboratory tests, as well as their changes from baseline will be statistically summarized by dose group and visit.
Clinical laboratory test: Hematology - eosinophil percentage | pre-dose, Day6, Day15, Day29, Day43, Day57
  The results of clinical laboratory tests, as well as their changes from baseline will be statistically summarized by dose group and visit.
Clinical laboratory test: Hematology - basophil count | pre-dose, Day6, Day15, Day29, Day43, Day57
  The results of clinical laboratory tests, as well as their changes from baseline will be statistically summarized by dose group and visit.
Clinical laboratory test: Hematology - basophil percentage | pre-dose, Day6, Day15, Day29, Day43, Day57
  The results of clinical laboratory tests, as well as their changes from baseline will be statistically summarized by dose group and visit.
Clinical laboratory test: Hematology - mean corpuscular hemoglobin (MCH) | pre-dose, Day6, Day15, Day29, Day43, Day57
  The results of clinical laboratory tests, as well as their changes from baseline will be statistically summarized by dose group and visit.
Clinical laboratory test: Hematology - mean corpuscular volume (MCV) | pre-dose, Day6, Day15, Day29, Day43, Day57
  The results of clinical laboratory tests, as well as their changes from baseline will be statistically summarized by dose group and visit.
Clinical laboratory test: Urinalysis | pre-dose, Day6, Day15, Day29, Day43, Day57
  Urine protein, cast, urine red blood cells, urine white blood cells, urine pH, urine ketone body, glucose urine, urine bilirubin, and urine occult blood
Clinical laboratory test: Biochemistry - Glucose (Glu) | pre-dose, Day6, Day15, Day29, Day43, Day57
  The results of clinical laboratory tests, as well as their changes from baseline will be statistically summarized by dose group and visit.
Clinical laboratory test: Biochemistry - alanine aminotransferase (ALT) | pre-dose, Day6, Day15, Day29, Day43, Day57
  The results of clinical laboratory tests, as well as their changes from baseline will be statistically summarized by dose group and visit.
Clinical laboratory test: Biochemistry - aspartate aminotransferase (AST) | pre-dose, Day6, Day15, Day29, Day43, Day57
  The results of clinical laboratory tests, as well as their changes from baseline will be statistically summarized by dose group and visit.
Clinical laboratory test: Biochemistry - alkaline phosphatase (ALP) | pre-dose, Day6, Day15, Day29, Day43, Day57
  The results of clinical laboratory tests, as well as their changes from baseline will be statistically summarized by dose group and visit.
Clinical laboratory test: Biochemistry - lactate dehydrogenase (LDH) | pre-dose, Day6, Day15, Day29, Day43, Day57
  The results of clinical laboratory tests, as well as their changes from baseline will be statistically summarized by dose group and visit.
Clinical laboratory test: Biochemistry - gamma-glutamyltransferase (γ-GGT) | pre-dose, Day6, Day15, Day29, Day43, Day57
  The results of clinical laboratory tests, as well as their changes from baseline will be statistically summarized by dose group and visit.
Clinical laboratory test: Biochemistry - serum total protein (TP) | pre-dose, Day6, Day15, Day29, Day43, Day57
  The results of clinical laboratory tests, as well as their changes from baseline will be statistically summarized by dose group and visit.
Clinical laboratory test: Biochemistry - albumin (ALB) | pre-dose, Day6, Day15, Day29, Day43, Day57
  The results of clinical laboratory tests, as well as their changes from baseline will be statistically summarized by dose group and visit.
Clinical laboratory test: Biochemistry - total bilirubin (TBIL) | pre-dose, Day6, Day15, Day29, Day43, Day57
  The results of clinical laboratory tests, as well as their changes from baseline will be statistically summarized by dose group and visit.
Clinical laboratory test: Biochemistry - direct bilirubin (DBIL) | pre-dose, Day6, Day15, Day29, Day43, Day57
  The results of clinical laboratory tests, as well as their changes from baseline will be statistically summarized by dose group and visit.
Clinical laboratory test: Biochemistry - blood urea nitrogen (BUN) | pre-dose, Day6, Day15, Day29, Day43, Day57
  The results of clinical laboratory tests, as well as their changes from baseline will be statistically summarized by dose group and visit.
Clinical laboratory test: Biochemistry - creatinine (Crea) | pre-dose, Day6, Day15, Day29, Day43, Day57
  The results of clinical laboratory tests, as well as their changes from baseline will be statistically summarized by dose group and visit.
Clinical laboratory test: Biochemistry - sodium (Na) | pre-dose, Day6, Day15, Day29, Day43, Day57
  The results of clinical laboratory tests, as well as their changes from baseline will be statistically summarized by dose group and visit.
Clinical laboratory test: Biochemistry - potassium (K) | pre-dose, Day6, Day15, Day29, Day43, Day57
  The results of clinical laboratory tests, as well as their changes from baseline will be statistically summarized by dose group and visit.
Clinical laboratory test: Biochemistry - chlorine (Cl) | pre-dose, Day6, Day15, Day29, Day43, Day57
  The results of clinical laboratory tests, as well as their changes from baseline will be statistically summarized by dose group and visit.
Clinical laboratory test: Biochemistry - calcium (Ca) | pre-dose, Day6, Day15, Day29, Day43, Day57
  The results of clinical laboratory tests, as well as their changes from baseline will be statistically summarized by dose group and visit.
Clinical laboratory test: Biochemistry - phosphorus (P) | pre-dose, Day6, Day15, Day29, Day43, Day57
  The results of clinical laboratory tests, as well as their changes from baseline will be statistically summarized by dose group and visit.
Clinical laboratory test: Biochemistry - triglycerides (TG) | pre-dose, Day6, Day15, Day29, Day43, Day57
  The results of clinical laboratory tests, as well as their changes from baseline will be statistically summarized by dose group and visit.
Clinical laboratory test: Biochemistry - total cholesterol (TC) | pre-dose, Day6, Day15, Day29, Day43, Day57
  The results of clinical laboratory tests, as well as their changes from baseline will be statistically summarized by dose group and visit.
Clinical laboratory test: Biochemistry - high-density lipoprotein cholesterol (HDL-C) | pre-dose, Day6, Day15, Day29, Day43, Day57
  The results of clinical laboratory tests, as well as their changes from baseline will be statistically summarized by dose group and visit.
Clinical laboratory test: Biochemistry - low-density lipoprotein cholesterol (LDL-C) | pre-dose, Day6, Day15, Day29, Day43, Day57
  The results of clinical laboratory tests, as well as their changes from baseline will be statistically summarized by dose group and visit.
Clinical laboratory test: Biochemistry - uric acid (UA) | pre-dose, Day6, Day15, Day29, Day43, Day57
  The results of clinical laboratory tests, as well as their changes from baseline will be statistically summarized by dose group and visit.
Clinical laboratory test: Biochemistry - creatine kinase (CK) | pre-dose, Day6, Day15, Day29, Day43, Day57
  The results of clinical laboratory tests, as well as their changes from baseline will be statistically summarized by dose group and visit.
Clinical laboratory test: Coagulation - International normalized ratio (INR) | pre-dose, Day6, Day15, Day29, Day43, Day57
  The results of clinical laboratory tests, as well as their changes from baseline will be statistically summarized by dose group and visit.
Clinical laboratory test: Coagulation - prothrombin time (PT) | pre-dose, Day6, Day15, Day29, Day43, Day57
  The results of clinical laboratory tests, as well as their changes from baseline will be statistically summarized by dose group and visit.
Clinical laboratory test: Coagulation - activated partial thromboplastin time (APTT) | pre-dose, Day6, Day15, Day29, Day43, Day57
  The results of clinical laboratory tests, as well as their changes from baseline will be statistically summarized by dose group and visit.
Clinical laboratory test: Coagulation - fibrinogen (FIB) | pre-dose, Day6, Day15, Day29, Day43, Day57
  The results of clinical laboratory tests, as well as their changes from baseline will be statistically summarized by dose group and visit.
Clinical laboratory test: Pregnancy test | pre-dose, Day15, Day29, Day43, Day57
  Blood pregnancy test (for females only)
Clinical laboratory test: Infectious serology | pre-dose
  Hepatitis B surface antigen, hepatitis B core antibody, hepatitis C antibody, Treponema pallidum antibody, and human immunodeficiency virus antibody
Clinical laboratory test: Blood alcohol test | pre-dose
  Blood alcohol test
Clinical laboratory test: Urine drug abuse screening | pre-dose
  Morphine, methamphetamine, ketamine, methylenedioxy methylamphetamine, marijuana, and cocaine
T-Spot | pre-dose
  If necessary, T-spot screening can be performed for priorly infected or suspected patients
Immunogenicity: The positive rate and titer of anti-drug antibody (ADA), and the positive rate of neutralizing antibody (Nab, in case of ADA positive results) | pre-dose, Day11, Day29, Day43, Day57
  Immunogenicity will be analyzed based on IMS. The number and percentage of subjects positive for CBP-201 ADA and Nab will be summarized by dose group.

CONTACTS AND LOCATIONS:
Overall Officials: Suzhou Connect, Study Director — Connect Biopharm LLC
Locations (1):
- The Second Hospital of Anhui Medical University, Hefei, Anhui, China